CLINICAL TRIAL: NCT06810804
Title: A Phase IIa Study to Evaluate the Efficacy and Safety of NBQ72S in Breast Cancer Patients With Leptomeningeal Metastases, With or Without Brain Parenchymal Metastases
Brief Title: A Phase IIa Study to Evaluate NBQ72S
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantong Bencao Quadriga Medical Technology Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBQ-72S-2001
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): All patients reated with NBQ72S
  Interventions: Drug: NBQ72S

INTERVENTIONS:
Drug: NBQ72S — Patients will receive the study drug every 28 days
  Other Names: QBS10072S

SUMMARY:
A phase IIa, single-arm, open-label study was conducted to evaluate the efficacy and safety of NBQ72S, in patients with leptomeningeal metastases from breast cancer. All patients will receive the study drug every 28 days until withdrawal from treatment.

DETAILED DESCRIPTION:
This is a single-arm, open-label study designed to evaluate the efficacy and safety of NBQ72S in patients with breast cancer leptomeningeal metastasis (with or without brain parenchymal metastasis).

Patients will undergo screening prior to study entry. After screening successfully, they will receive intravenous infusion of NBQ72S. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of informed consent, or any other conditions except as specified in the protocol (whichever occurs first). However, patients who demonstrate clinical benefits (despite radiological progression) with manageable toxicity, and are willing to continue receiving the NBQ72S, will be given the opportunity to continue treatment after the assessment and confirmation of Investigator.

After treatment completion, patients will undergo safety follow-up and long-term survival follow-up until death or lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have histological evidence confirming the diagnosis of breast cancer with leptomeningeal metastasis: a. Breast cancer must be diagnosed through biopsy from either the primary or metastatic sites; b. Leptomeningeal metastasis (with or without brain parenchymal metastases) must be confirmed by imaging examinations(MRI), or by positive or suspicious cerebrospinal fluid cytology; c. There is no restriction on the duration of prior systemic therapy for the primary tumor.
* The patient's Karnofsky Performance Status (KPS) must be ≥60.
* The patient must have adequate bone marrow function, including:

  1. Absolute neutrophil count (ANC) ≥1,500/mm³ or ≥1.5 x 10⁹/L;
  2. Platelet count ≥100,000/mm³ or ≥100 x 10⁹/L;
  3. Hemoglobin ≥9 g/dL;
* The patient must have adequate renal function, including:

  a. Serum creatinine ≤1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥50 mL/min. Note: In equivocal cases, a 24-hour urine collection test can be used to estimate the creatinine clearance more accurately;
* The patient must have adequate hepatic function, including:

  1. Total serum bilirubin ≤1.5 x ULN; if the tumor involves the liver, or if the patient has a history of Gilbert's syndrome, total bilirubin must be <3 x ULN;
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN; if the tumor involves the liver, these values must be ≤5.0 x ULN;
* Females of childbearing potential and males with fertile partners must agree to use effective contraception during the study and for 7 months following the last dose of study treatment;

Exclusion Criteria:

* Patients with any other active malignancies unrelated to the primary tumor, except for those with basal cell carcinoma, squamous cell carcinoma, or in situ carcinoma that have been adequately treated.
* Patients who are intolerant to any substance in the investigational product, including sulfobutylether-β-cyclodextrin, mefenamic acid, bendamustine, chloramphenicol, or any nitrogen mustard chemotherapy agents, or who have experienced a severe (Grade ≥3) allergic or hypersensitivity reaction to these substances.
* Patients who have received a live vaccine or experimental drug within 30 days prior to Cycle 1, Day 1 (C1D1).
* Pregnant or breastfeeding patients.
* Any other conditions that may affect the patient's eligibility for this study in the judgment of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
OS | through study completion, an average of 1.5 years
  Overall Survival

SECONDARY OUTCOMES:
Intracrarnial PFS | through study completion, an average of 1.5 years
  Intracrarnial Progression Free Survival
Intracrarnial DOR | through study completion, an average of 1.5 years
  Intracrarnial Duration of Response
Extracrarnial ORR | through study completion, an average of 1.5 years
  Extracrarnial Objective Response Rate
Extracrarnial PFS | through study completion, an average of 1.5 years
  Extracrarnial Progression Free Survival
Extracrarnial DOR | through study completion, an average of 1.5 years
  Extracrarnial Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No